CLINICAL TRIAL: NCT05487755
Title: Investigational and Comparative Study to Assess Safety and Effectiveness of Tadalafil and Pentoxifyllin in the Management of Diabetic Nephropathy
Brief Title: Investigational and Comparative Study in the Management of Diabetic Nephropathy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Walla Ahmed Amaar, clinical pharmacist, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DN mangement
Record Dates: First submitted 2022-07-22; First posted 2022-08-04 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Diabetic Nephropathy Type 2
MeSH Terms: interventions — Tadalafil; Tablets; Pentoxifylline

STUDY DESIGN:
Intervention Model Description: * This is a randomized, controlled, prospective study.
  * Ninety diabetic nephropathy patients at stage 3(micro-albuminuria) will be divided into three groups as follow -Group 1: (n=30) control group will receive traditional therapy blood glucose lowering agent +RAAS blockade ACEI or ARBs for six months.
    * Group 2 :( n=30) will receive traditional therapy +tadalafil PO 20 mg every other day for six months.
  Group 3 :( n=30) will receive traditional therapy+ pentoxifylline PO 400 mg twice daily for six months.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (No Intervention): : (n=30) control group will receive traditional therapy blood glucose lowering agent +RAAS blockade ACEI or ARBs for six months.
- Tadalafil group (Experimental): :( n=30) will receive traditional therapy +tadalafil PO 20 mg every other day for six months
  Interventions: Drug: Tadalafil 20Mg Oral Tablet
- pentoxifylline group (Experimental): :( n=30) will receive traditional therapy+ pentoxifylline PO 400 mg twice daily for six months.
  Interventions: Drug: Pentoxifylline 400 MG Oral Tablet

INTERVENTIONS:
Drug: Tadalafil 20Mg Oral Tablet — Tadalafil is a phosphodiesterase type 5 enzyme (PDE5) inhibitor used mainly in erectile dysfunction and pulmonary hypertension by a mechanism involving increase(NO-cGMP-PKG) signaling pathway.(8) Tadalafil is a powerful pleiotropic drug that it can be used in DN as it can target more than pathway involved in pathogenesis of DN include hyperglycemia and endothelial dysfunction through increase (NO-cGMP) signaling pathway as well as hyperlipidemia
  Other Names: cialong
  Arms: Tadalafil group
Drug: Pentoxifylline 400 MG Oral Tablet — Pentoxifylline is a methyl xanthine derivative, non selective phosphodiesterase enzyme inhibitor used mainly to treat peripheral vascular diseases by improve blood flow
  Other Names: Pental SR
  Arms: pentoxifylline group

SUMMARY:
The objective of this study is to investigate and compare the safety and efficacy of selective (PDE5) enzyme inhibitor; tadalafil and non selective (PDE) inhibitor; pentoxifylline in diabetic nephropathy to improve glucose metabolism, lipid profile and decrease albuminuria.

DETAILED DESCRIPTION:
Diabetic nephropathy(DN) is one of the major micro- vascular complications of diabetes mellitus and the leading cause of end-stage renal disease (ESRD) that require renal replacement therapies.

The average incidence of diabetic nephropathy is 3% per year during the first 10 to 20 years after diabetes onset. Diabetic nephropathy occurs in 20-40% of all diabetic patients.

Pathogenesis of diabetic nephropathy is complex and multi-factorial in which diabetes mellitus has more than pathway for initiation and progression of the disease.

* Metabolic pathway: result in formation of advanced glycation end products (AGEs).
* Inflammatory pathway: result in increase serum level of tumor necrosis factor-α(TNF .
* Hemodynamic pathway: result in increase serum level of endothelin-1 which result in glomerular hypertension and hyper filtration.

Tadalafil is a phosphodiesterase type 5 enzyme (PDE5) inhibitor used mainly in erectile dysfunction and pulmonary hypertension by a mechanism involving increase(NO-cGMP-PKG) signaling pathway.

Tadalafil is a powerful pleiotropic drug that it can be used in DN as it can target more than pathway involved in pathogenesis of DN include hyperglycemia and endothelial dysfunction through increase (NO-cGMP) signaling pathway as well as hyperlipidemia. Animal studies reported that tadalafil increase significantly total antioxidant capacity(TAC),decrease significantly serum level of inflammatory marker (TNF- α), blood glucose level, serum creatinine ,serum urea and urinary albumin excretion all result in decrease renal inflammation, injury, necrosis and apoptosis.

Pentoxifylline is a methyl xanthine derivative, non selective phosphodiesterase enzyme inhibitor used mainly to treat peripheral vascular diseases by improve blood flow, increase red blood cell flexibility and inhibit platelet aggregation.

Pentoxifylline have been recently widely used in many animal studies and clinical trials to evaluate its efficacy in management of DN and the results were so promising.(14)

Pentoxifylline can slow the decrease in eGFR, and significantly reduce albuminuria in which it can be effective alternative to ACEI in reducing albuminuria as proved by clinical trial.(15) The powerful effect of pentoxifylline in DN as it can affect several pathways implicated in pathogenesis of DN; it has hypoglycemic effect by decrease Significantly blood glucose, HbA1c and serum triglyceride, it also decrease pro inflammatory cytokines (TNF-α, IL-1, IL-6), reduce plasma level of malondialdehyde and increase glutathione level.(16)

Neutrophil Gelatinase-Associated Lipocalin (NGAL): is a 25-kDa protein belong to lipocalin superfamily. The urinary concentration of NGAL increase in renal tubular damage as a result of both diminished reabsorption and increased release from renal tubules into urine indicating both proximal and distal tubular damage respectively.(17) NGAL is not considered a marker of renal function but a marker of structural damage of renal tubules, its level can quantify the degree of tubular damage.(18) NGAL can be used as a precocious marker of therapeutic response by application of NGAL measurement in monitoring the effectiveness of a particular treatment and predicting different clinical outcomes in the course of renal diseases

ELIGIBILITY:
Inclusion Criteria:

* A confirmed with clinical diagnosis of T2DM with duration at least 7 years to ensure established of micro-vascular complication (DKD).
* females (post-menopause), males with sufficient erectile function.
* Patients on stage 3 DN with evidence of persistent micro-albuminuria. All Abnormal tests of (UACR) must be confirmed in two out of three samples collected over a 6 month period before enrolled in the study.
* (urinary ACR≥30-300mg/g) in 3 consecutive measurements in 6 months period despite treatment with RAAS blockade(ramipril 10 mg ) ACEI or for at least 6 months period before enrollment in the study at maximum recommended tolerated dose.

Exclusion Criteria:Cardiovascular disease: angina, arrhythmias, myocardial Infarction, heart failure (NYHA II -IV), uncontrolled hypertension > (170 \100 mm Hg) severe hypotension < (90\50 mm Hg), Hearing problem, vision defect, previous episodes of retinal / cerebral hemorrhage, psychiatric disease, thyroid disorders, alcohol abuse, smoking, Hepatic insufficiency (child -Pugh class C), (ALT or AST>3N), cholestasis, history of chronic inflammatory, immunologic or malignant disease. Acute inflammation or infectious disease in the previous 3 months, taking immunosuppressive treatment, Known allergy to tadalafil or methylxanthine, Use alpha one blockers, use of anti-oxidant drugs three months before enrollment in the study ,medications strongly alter CYP3A4 inducer or inhibitor, use of nitrates, other PDEI drugs, - Renal disease (acute kidney injury, recent exposure to radio- contrast media, creatinine clearance <30 ml/ min /1.73 m2 , bleeding disorders, peptic ulcer, and stroke, Pregnancy, lactation.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Change in Urinary albumin/creatinine ratio (ACR) | Change between baseline and six months after
  Measurement of urine albumin to creatinne ratio by measurement of urine albumin using Turbidimetric immunoassay method and measurement of urine creatinnie by standard by enzymatic colorimetric methods
Change in Hemoglobin A1c (HbA1c). | Change between baseline and six months after
  Measurement of Hemoglobin A1C using (HPLC: ion exchange chromatography)
Change in Fasting blood glucose. | Change between baseline and six months after
  Measurement of Fasting blood glucose by using standard enzymatic colorimetric methods
Change in Sr Cr | Change between baseline and six months after
  Measurement of serum creatinine using colorimetric technique
Change in Creatinine clearance | Change between baseline and six months after
  Creatinine clearance was calculated by (Cockcroft-Gault Formula)
change in 2- Hours Postprandial blood glucose | Change between baseline and six months after
  Measurement 2- Hours Postprandial blood glucose in blood using standard enzymatic colorimetric methods

SECONDARY OUTCOMES:
Change in serum ((TNF-α). | Change between baseline and six months after
  Measurement of serum level of (TNF-α) by Enzyme linked immunosorbent assay (ELISA).
Change in Urinary NGAL (uNGAL). | Change between baseline and six months after
  Measurement of urinary Neutrophil Gelatinase-Associated Lipocalin (NGAL)using by Enzyme linked immunosorbent assay ELISA technique:
Change in Lipid profile (TG, LDL, and HDL). | Change between baseline and six months after
  Measurement of serum lipid profile (TC,TG,HDL,LDL)using Enzymatic Colorimetric Method
Change in serum malondialdehyde (MDA) . | Change between baseline and six months after
  Meaurement of serum malondialdehyde by Enzyme linked immunosorbent assay (ELISA) .

CONTACTS AND LOCATIONS:
Overall Officials: Wafaa S Hegab, Lecturer, Study Chair — Tanta University
Locations (1):
- Faculty of pharmacy, Tanta, Egypt

REFERENCES:
- [Background] Rivero A, Mora C, Muros M, Garcia J, Herrera H, Navarro-Gonzalez JF. Pathogenic perspectives for the role of inflammation in diabetic nephropathy. Clin Sci (Lond). 2009 Mar;116(6):479-92. doi: 10.1042/CS20080394. PMID 19200057
- [Background] Wada J, Makino H. Inflammation and the pathogenesis of diabetic nephropathy. Clin Sci (Lond). 2013 Feb;124(3):139-52. doi: 10.1042/CS20120198. PMID 23075333
- [Derived] Hegazy SK, Amaar WA, Hegab WSM. Tadalafil versus pentoxifylline in the management of diabetic kidney disease: a randomized clinical trial. Diabetol Metab Syndr. 2024 Jun 24;16(1):138. doi: 10.1186/s13098-024-01363-3. PMID 38915115